CLINICAL TRIAL: NCT02807311
Title: OPTIMIZATION OF NUTRITIONAL MANAGEMENT OF PATIENTS WAITING FOR LUNG TRANSPLANT INTO Strasbourg University Hospitals
Acronym: nONsTOP
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6369
Record Dates: First submitted 2016-06-15; First posted 2016-06-21 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2016-05

CONDITIONS: Malnutrition
Keywords: Malnutrition; Undernutrition; lung transplantation; artificial nutrition; nutritional supplements; enteral nutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Undernutrition is the result of energy and protein deficiency and / or catabolic. These phenomena are observed daily in patients awaiting lung transplantation.

After lung transplantation that undernutrition is growing (on average 11% weight loss after the first observations in the continuing care of the University Hospital of Strasbourg). In other words the non-malnourished patients become. Hence the importance to reach every patient awaiting transplant, mainly to patients already malnourished before surgery.

Several studies have shown that early nutritional support has a direct effect on reducing comorbidities and the average length of stay. In the course of care of these patients it is necessary to intensify the dietary management to give them the best chance for early rehabilitation.

The main objective of the study is to evaluate the impact of the use of the SFNEP's nutritional care decision-making tree (Société Francophone Nutrition Clinique et Métabolisme) on the implementation of enteral nutrition by gastrostomy tube in patients awaiting for lung transplantation.

ELIGIBILITY:
Inclusion criteria:

transplant patients between January 1, 2012 and December 31, 2015 aged over 16 years, with a BMI <25 at the time of pre-transplant assessment and that not oppose the use of his data.

Exclusion criteria:

* Cardiopulmonary Transplant Patients
* refusal to participate in the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: transplant patients between January 1, 2012 and December 31, 2015 aged over 16 years, with a BMI <25 at the time of pre-transplant assessment
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2016-08-17 (Actual); Primary Completion 2016-08-22 (Actual); Study Completion 2017-02-16 (Actual)

PRIMARY OUTCOMES:
Assessment of the proportion undernourished patients by using the SFNEP's nutritional care decision-making tree | befor pulmonary transplantation, up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sophie BOURA, Dietician, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Service de pneumologie - Nouvel Hôpital Civil, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No